CLINICAL TRIAL: NCT00002168
Title: An Open Label, Randomized, Comparative Study of Zerit (d4T) + Videx (ddI) + Crixivan Versus Retrovir (AZT) + Epivir (3TC) + Crixivan in HIV-Infected, Antiretroviral Naive Subjects With CD4 Cell Counts of 200 - 700/mm3 and HIV RNA Baseline Copy Number of >= 10,000 Copies/ml
Brief Title: A Comparison of Two Anti-HIV Triple-Drug Combinations in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 260B; BMS 002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Zidovudine; Stavudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Lamivudine; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two anti-HIV drug combinations when given to HIV-infected patients who have never been treated with anti-HIV drugs. One drug combination is stavudine (d4T) plus didanosine (ddI) plus Crixivan. The other combination is Retrovir (AZT) plus Epivir (3TC) plus Crixivan.

DETAILED DESCRIPTION:
100 patients will be randomized to receive Zerit (Stavudine) + Videx (Didanosine) + Crixivan (Indinavir) and 100 patients will be randomized to receive Retrovir (Zidovudine) + Epivir (Lamivudine) + Crixivan (Indinavir).

Patients will be treated for 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 cell count of 200 - 700 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

AIDS defining condition within 1 month of study entry.

Prior Medication:

Excluded:

Patients with any history of antiretroviral therapy treatment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - East Bay AIDS Clinic, Berkeley, California
  - Harbor UCLA Med Ctr / Division of Immunology / N-24, Torrance, California
  - Anderson Clinical Research, Washington D.C., District of Columbia
  - George Washington Med Ctr / Clinical Trials Unit, Washington D.C., District of Columbia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Northwestern Univ, Chicago, Illinois
  - Univ of Nebraska, Omaha, Nebraska
  - Univ of North Carolina / Infectious Disease Division, Chapel Hill, North Carolina
  - The Nalle Clinic / Clinical Research Dept, Charlotte, North Carolina
  - Univ of Pennsylvania / Infectious Diseases Division, Philadelphia, Pennsylvania
  - Southwest Infectious Disease Association / PA, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
- Hosp Regional de Ponce - Area Vieja, Ponce, Puerto Rico